CLINICAL TRIAL: NCT04269512
Title: Prospective Randomized Trial to Evaluate the Prognostic Role of Lymphnode Dissection in Men With Prostate Cancer Treated With Radical Prostatectomy (Predict-Study)
Brief Title: Role of Lymphnode Dissection in Men With Prostate Cancer Treated With Radical Prostatectomy
Acronym: PREDICT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDICT_MK2019
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; lymphadenectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extended lymph node dissection (Active Comparator): Patients randomized to arm A undergo bilateral lymph node dissection in the pelvic area as part of prostatectomy. At least 10 lymph nodes must be removed.
  Interventions: Procedure: lymph node dissection
- standard without lymph node dissection (No Intervention): Application of standardized surgical technique without extensive lymph node dissection. If, contrary to expectation, intraoperative suspicion of lymphogenic metastasis results, a lymph node dissection is performed and the patient is excluded from the study (freedom of the surgeon).

INTERVENTIONS:
Procedure: lymph node dissection — At least 10 lymph nodes must be removed.
  Arms: extended lymph node dissection

SUMMARY:
Currently, lymph node dissection is standard of care during prostatectomy of intermediate risk tumors at the Martini Clinic. It allows the assessment of possible but unlikely lymph nodes metastases. In case of lymph node metastasis, depending on the number of affected lymph nodes, an adjuvant radiation with or without additional hormone therapy may be discussed in order to stop or delay further progression of the disease.

Since the procedure carries additional risks, it is controversial. The risks include prolonged surgery duration, injury of vessels and nerves, as well as disorders of lymphatic circulation after surgery. Moreover, formation of lymphoceles (accumulation of lymph fluid in the tissue) are common, which may result in soft tissue swelling, thrombosis, inflammation and additional surgical procedures.

Therefore, the aim of this study is to evaluate whether the removal of the lymph nodes during prostatectomy positively influences the course of the disease in patients with intermediate risk prostate cancer, or if the lymph node dissection does not have any influence on the recurrence of the disease and therefore further therapies.

In this case, the omission of lymph node dissection may avoid an unnecessary expansion of the operation and the potentially associated side effects linked to it. This is particularly of interest considering the rapidly advancing technical possibilities, both in imaging and in the treatment of prostate cancer, since this enables an earlier and more individual intervention in the case of recurrence.

DETAILED DESCRIPTION:
The significance of lymph node dissection in radical prostatectomy has not been conclusively clarified. If a radical prostatectomy is planned, the question occurs if the additional pelvic lymph node dissection (LND) is justified and to what extent it should be performed (limited LND, standard LND or extended LND). On the one hand, the detection of lymph node metastases is associated with a significantly worse course of the tumor disease and requires immediate or delayed hormone-ablative therapy. On the other hand, the lymph node dissection is associated with risks (lymphoceles, thromboses, lymphedema), so that the indication in negative lymph node findings appears questionable. It must be weighed between the diagnostic advantage and the possibility of increased morbidity due to the lymphadenectomy. For localized intermediate risk prostate cancer (PSA> 10 ng / ml - 20 ng / ml or Gleason score 7 or cT category 2b ), there are currently no recommendations for performing a lymph node dissection during prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* localized intermediate risk prostate cancer (intermediate risk (PSA> 10 ng / ml - 20 ng / ml or Gleason score 7 or cT category 2b)
* scheduled for open radical prostatectomie or DaVinci prostatectomie

Exclusion Criteria:

* American Society of Anesthesiology Classification> 3
* Existing contraindications for performing a lymph node dissection
* Neoadjuvant hormone therapy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Enrollment: 3650 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
PSA recurrence rate | 36 months after surgery
  The PSA recurrence rate in patients with intermediate risk prostate cancer treated with radical prostatectomy with or without additional lymph node dissection at three years of follow up (PSA recurrence: PSA value ≥ 0.2 ng / ml).

SECONDARY OUTCOMES:
Incidence of lymphoceles and complications | 6 months after surgery
  (Clavien classification)
quality of life including continence and potency | 6, 12, 24, 36 months after surgery
  Questionnaire Expanded prostate cancer index composite (EPIC-26)
metastasis-free survival | 36 months
  diagnosis of metastasis after prostatectomy by radiological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Markus Graefen, Principal Investigator — Director
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Homepage — http://www.martini-klinik.de